CLINICAL TRIAL: NCT03497819
Title: Pilot Study of Autologous Chimeric Antigen Receptor Cells Against Mesothelin and CD19 in Patients With Pancreatic Cancer
Brief Title: Autologous CARTmeso/19 Against Pancreatic Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Meng-Tao Zhou, Director, First Affiliated Hospital of Wenzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YXA-meso19
Record Dates: First submitted 2017-10-27; First posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Pancreatic Cancer
Keywords: CART; Pancreatic Cancer; artery infusion
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CARTmeso/19 treatment arm (Experimental): Patients with pancreatic cancer receiving CARTmeso and CART19 autologous cells via artery infusion or i.v. with cyclophosphamide precondition
  Interventions: Biological: CARTmeso CART19

INTERVENTIONS:
Biological: CARTmeso CART19 — Autologous chimeric antigen receptor T cells with murine scFv, 41BB co-stimulatory domain and CD3ζ signaling domain targeting mesothelin or CD19

SUMMARY:
Pancreatic cancer patients receive chimeric antigen receptor (CAR) T cells against mesothelin (CARTmeso) or CD19 (CART19) cells administered at 3 days via pancreatic artery infusion or i.v. after preconditioning of cyclophosphamide. Both CART cells are autologous. CARTmeso cells target pancreatic cells which highly express mesothelin, while CART19 cells target tumor-associated B cells expressing cluster of differentiation antigen 19 (CD19) which are mostly immunosuppressive. The investigators hypothesize that this combination therapy may enhance the efficacy of CARTmeso cells in the body. Additionally, a medium dose of cyclophosphamide is used to enhance the engraftment of CART cells.

DETAILED DESCRIPTION:
This is a single arm, open-label, pilot study to determine the safety and feasibility of combination CARTmeso cells and CART19 cells in patients with pancreatic cancer following lymphodepletion with cyclophosphamide. Both cells contain CAR proteins consisting of a murine-derived single chain antibody fragment (scFv), cluster of differentiation antigen 137 (41BB) co-stimulatory domain and cluster of differentiation antigen 3 zeta chain (CD3ζ) signaling domain transduced by lentivirus

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* serum soluble mesothelin-related protein (SMRP) > 0.4 nanomolar/L
* Persistent cancer after at least one prior standard of care chemotherapy for advanced stage disease

  * 18 years of age and ≤65
* Life expectancy greater than 3 months
* Satisfactory organ and bone marrow function

Exclusion Criteria:

* Participation in a therapeutic investigational study within 4 weeks prior to the screening visit
* Active invasive cancer other than pancreatic cancer
* HIV, hepatitis B/C virus, or infections
* Active autoimmune disease requiring immunosuppressive therapy within 4 weeks
* Planned concurrent treatment with systemic high dose corticosteroids
* Patients requiring supplemental oxygen therapy
* Pregnant or breastfeeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
The Percentage of Adverse Events (AEs) ≥ grade 3 assessed through MedDra and CTCAE v4.03 [Time frame: from infusion to 3 month afterward] | From first infusion to 3 months afterward
  Primary outcome is the percentage of adverse events (AEs) ≥ grade 3. AEs are assessed through MedDra and CTCAE v4.03. Any patients who receive any dose of CART cells will be evaluated

SECONDARY OUTCOMES:
Overall Response Rate defined as any improvement measured by imaging following RECIST 1.1 [Time Frame: Day 14 and 1 month after infusion] | Day 14 and 1 month after infusion, or until patient withdraw consent or receive new therapy
  Secondary outcome is overall response rate. A response is defined as any improvement measured by imaging following RECIST 1.1. Only patients who receive infusions per protocol will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Mengtao Zhou, MD, Principal Investigator — First Affiliated Hospital of Wenzhou Medical University
Locations (1):
- First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No